CLINICAL TRIAL: NCT00060996
Title: A Randomized Placebo-Controlled, 12-Week Multicenter Study of the Safety and Efficacy of Continuous or Daily Administration of Remodulin® (Treprostinil Sodium) Injection in Patients With CLI With No Planned Revascularization Procedures
Brief Title: Study of Remodulin in Patients With Critical Limb Ischemia With No Planned Revascularization Procedures
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REM 03:202
Record Dates: First submitted 2003-05-19; First posted 2003-05-20 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Critical Limb Ischemia; Peripheral Vascular Disease; Foot Ulcers; Rest Leg Pain
Keywords: Critical Limb Ischemia; Peripheral Vascular Disease; UT-15; Remodulin; treprostinil
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Peripheral Vascular Diseases; Foot Ulcer | interventions — treprostinil; Injections

INTERVENTIONS:
Drug: Remodulin® (treprostinil sodium) Injection

SUMMARY:
The purpose of this study is to assess and compare the safety of continuous and daily subcutaneous Remodulin therapy in patients with critical limb ischemia (CLI) with no planned vascular interventional procedures; and to determine the effect of Remodulin on wound healing and treadmill walk distance.

ELIGIBILITY:
Patients with Stage III or IV critical limb ischemia due to documented peripheral arterial disease with no planned interventional vascular procedures

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2003-02; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wade, PhD, Study Director — United Therapeutics
Locations (7):
- United States (7):
  - University of South Florida College of Medicine, Tampa, Florida
  - University of Massachusetts Memorial Health, Worcester, Massachusetts
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Oregon Health Sciences University, Portland, Oregon
  - Presbyterian Medical Center, Philadelphia Heart Institute, Philadelphia, Pennsylvania
  - South Carolina Heart Center, Columbia, South Carolina
  - The Methodist Hospital, Houston, Texas